CLINICAL TRIAL: NCT01023347
Title: A Trial of Paclitaxel (Genexol®) and Cisplatin Versus Paclitaxel Loaded Polymeric Micelle (Genexol-PM®) and Cisplatin in Advanced Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samyang Biopharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GPM-0801
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; genexol-PM

ARMS (2):
- Paclitaxel (Genexol®) and Cisplatin (Active Comparator)
  Interventions: Drug: Paclitaxel (Genexol®)
- Paclitaxel loaded polymeric micelle (Genexol-PM®) & Cisplatin (Experimental)
  Interventions: Drug: Paclitaxel loaded polymeric micelle (Genexol-PM®)

INTERVENTIONS:
Drug: Paclitaxel (Genexol®)
  Arms: Paclitaxel (Genexol®) and Cisplatin
Drug: Paclitaxel loaded polymeric micelle (Genexol-PM®)
  Arms: Paclitaxel loaded polymeric micelle (Genexol-PM®) & Cisplatin

SUMMARY:
This is a randomized clinical trial of Paclitaxel (Genexol®) and Cisplatin versus Paclitaxel loaded polymeric micelle (Genexol-PM®) and Cisplatin in advanced non small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological evidence of locally advanced, metastatic or recurrent NSCLC (stage IIIB or Iv)
* At least one measurable lesion(s) by RECIST criteria
* No previous palliative chemotherapy
* Age 18 or higher.
* ECOG PS 0-2
* Life expectancy of at least 3 months.
* Adequate hematologic, hepatic, renal function
* Adequate bone marrow function (≥ ANC 1,500/ul, ≥ platelet 100,000/ul)
* Adequate liver function (≤ Total bilirubin ≤ 1.5 upper normal limit, ≤ AST/ALT x 2.5 upper normal limit, Alkaline phosphatase ≤ 2.5 upper normal limit)
* Adequate renal function (≤ serum creatinine 1.5 mg/dl)
* Written informed consent

Exclusion Criteria:

* No prior chemotherapy for NSCLC
* Patients with malignancies (other than NSCLC), except for adequately treated nonmelanoma skin cancer or in situ carcinoma of the cervix.
* Peripheral neuropathy ≥ grade 2 (NCI CTC, version 3.0)
* Clinically significant cardiac disease (medically uncontrollable heart disease)
* Active infection or other serious medical illness
* Contraindication to any drug contained in the chemotherapy regimen
* Pregnant or lactating women were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2008-06 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
response rate | up to 6 cycles
  overall responses are complete response and partial response

SECONDARY OUTCOMES:
overall survival | up to 3 years
  OS was calculated by the time from randomization date to the date of death
progression-free survival | up to 3 years
  PFS was calculated by the time from randomization date to objective tumor progression or death.
toxicity profiles | up to 6 cycles
  Incidence of AE, laboratory test results (hematology, blood chemistry, and urine test), physical examination, vital sign, and ECOG performance were used for safety endpoints

CONTACTS AND LOCATIONS:
Overall Officials: Sun Young Kim, Ph.D., Principal Investigator — Chungnam National University Hospital
Locations (1):
- Chungnam National University Hospital, Daejeon, Jung-gu, South Korea